CLINICAL TRIAL: NCT05316519
Title: Transcutaneous Auricular Vagus Nerve Stimulation: Mechanisms and Therapeutic Potential
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation to Enhance Motor Learning
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Pilot protocol terminated to begin trial.
Sponsor: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael A. Urbin, Scientist, VA Pittsburgh Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1619399
Record Dates: First submitted 2022-03-16; First posted 2022-04-07 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Neurological Injury; Motor Disorders; Paresis
MeSH Terms: conditions — Trauma, Nervous System; Motor Disorders; Paresis

STUDY DESIGN:
Intervention Model Description: Sham-controlled
Who Masked: Participant
Masking Description: Single-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous Vagus Nerve Stimulation (Experimental): Transcutaneous vagus nerve stimulation paired with visuomotor task training
  Interventions: Other: Transcutaneous Vagus Nerve Stimulation
- Transcutaneous Stimulation (Sham) (Placebo Comparator): Transcutaneous stimulation paired with visuomotor task training
  Interventions: Other: Transcutaneous Vagus Nerve Stimulation

INTERVENTIONS:
Other: Transcutaneous Vagus Nerve Stimulation — Visuomotor task training with transcutaneous stimulation targeting landmark that activates biomarker

SUMMARY:
Vagus nerve stimulation (VNS) activates neural pathways leading to the release of chemicals that promote plasticity and learning. Previous work has shown that the auricular branch of the vagus nerve innervates landmarks on the external ear. Work from the PI's laboratory has shown that electrical current applied to the external ear activates neural pathways implicated in the therapeutic effects of VNS. The broad objective of this project is to better understand physiological mechanisms that are modulated by auricular stimulation and its potential to enhance motor learning.

ELIGIBILITY:
Inclusion Criteria:

(For prospective subjects diagnosed with stroke)

* Confirmed diagnosis of a single stroke at least six months prior to participation

Exclusion Criteria:

* History of vestibular disorders or dizziness
* Diagnosis of neurological disorders affecting movement
* Ocular disease and/or impairment in more than one eye
* Pregnant or expecting to become pregnant
* Difficulty maintaining alertness and/or remaining still

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Precision grip stability (coefficient of variation or root-mean-square error) | 1 month post training
  The ability to stabilize precision grip according to target force and/or preload force will be quantified by calculating coefficient of variation (CV) or root-mean-square error (RMSE) which characterize variability in relation to mean force or target force.

SECONDARY OUTCOMES:
Force signal composition (Fourier transform) | 1 month post training
  The force signal oscillates at various frequencies and will be decomposed with a Fourier transform to quantify the relative contribution of higher frequencies.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Engineering Research Laboratories, Pittsburgh, Pennsylvania, United States